CLINICAL TRIAL: NCT03778008
Title: Recombinant Bovine Basic Fibroblast Growth Factor for the Treatment of Radiation Induced Oral Mucositis：An Open, Randomized, Controlled, Prospective Study
Brief Title: Recombinant Bovine Basic Fibroblast Growth Factor for the Treatment of Radiation Induced Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL003
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Stomatitis
Keywords: Radiation therapy; Nasopharyngeal carcinoma
MeSH Terms: conditions — Stomatitis; Nasopharyngeal Carcinoma | interventions — Gentamicins; Vitamin B 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant bovine basic fibroblast growth factor (Experimental)
  Interventions: Drug: Recombinant bovine basic fibroblast growth factor
- Quadruple mixture (Active Comparator): Quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and lidocaine composition
  Interventions: Combination Product: Quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and lidocaine composition

INTERVENTIONS:
Drug: Recombinant bovine basic fibroblast growth factor — Recombinant bovine basic fibroblast growth factor is prescribed at the beginning of radiotherapy for free. Patients are asked to start application of recombinant bovine basic fibroblast growth factor at the onset of radiotherapy, four times a day (after meals and before bedtime), until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation-induced oral mucositis. When grade > 3 OM happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted.
  Arms: Recombinant bovine basic fibroblast growth factor
Combination Product: Quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and lidocaine composition — Quadruple mixture is prescribed at the beginning of radiotherapy. Patients are asked to start application of quadruple mixture at the onset of radiotherapy, four times a day (before meals and before bedtime), until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation-induced oral mucositis. When grade > 3 OM happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted.
  Arms: Quadruple mixture

SUMMARY:
Radiation therapy is one of the treatments for Nasopharyngeal carcinoma . The most common side effects of post-radiation may be radiation-induced oral mucositis . When severe, oral mucositis increases the risk of infection and may affect clinical outcomes due to treatment interruption, dose reduction, and reduced treatment compliance. In China, a quadruple mixture of dexamethasone, gentamicin, vitamin B12, and lidocaine is commonly used in patients who begin to have radiation-induced oral mucositis . However, the incidence of radiation-induced oral mucositis remains high. Recombinant bovine basic fibroblast growth factor is a multifunctional cell growth factor that stimulates the growth of cells derived from mesoderm and neuroectodermal cells and thus has a wide range of biological activities. The drug has different degrees of promotion on the three stages of the wound repair process, namely the local inflammatory reaction stage, cell proliferation and differentiation, granulation tissue formation stage and tissue reconstruction stage. The purpose of this randomized controlled trial was to evaluate the efficacy of recombinant bovine basic fibroblast growth factor as an intervention in radiation-induced oral mucositis for the treatment of nasopharyngeal carcinoma , with a commonly used quadruple mixture (from dexamethasone, gentamicin , vitamin B12 and lidocaine composition) were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed and previously untreated nasopharyngeal carcinoma
2. Age ≥ 18 years and ≤ 65 years.
3. Karnofsky performance status (KPS) score ≥ 70
4. Planned to receive radiotherapy alone or concurrent chemoradiotherapy
5. Adequate bone marrow function: while blood cell >= 3,000/μL, absolute neutrophil count >= 1,500/μL, hemoglobin >= 100g/L, platelet >= 75,000/μL.
6. Life expectancy of >= 3 months.

Exclusion Criteria:

1. Younger than 18 years old or older than 70 years old
2. Pregnancy or lactation
3. Severe cerebrovascular disease/canker/psychosis/uncontrolled diabetes
4. Have suffered from oral diseases or salivary gland diseases or mow suffering from oral diseases or salivary gland diseases
5. Refuse to give up smoking/drinking/betel chewing
6. suffering from other active infection diseases and in need of treatment.
7. Known allergic reaction to any component of Recombinant Bovine Basic Fibroblast Growth Factoor or quadruple mixture, which is composed of dexamethasone, gentamicin, vitamin B12, and lidocaine, or severe allergic constitution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-21 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 mucositis | Day 56 after completion or termination of radiotherapy
  Incidence of grade ≥ 3 mucositis according to CTCAE version 5.0
EORTC QLQ-C30 | Day 56 after completion or termination of radiotherapy
  EORTC QLQ-C30 is a Quality-of-Life Instrument proposed by the European Organization for Research and Treatment of Cancer (EORTC), for use in International Clinical Trials in Oncology. The QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.
WHO score | Day 56 after completion or termination of radiotherapy
  The World Health Organization (WHO) Oral Toxicity score combines both elements into a single score that grades the severity of the condition from 0 (no oral mucositis) to 4 (swallowing not possible such that patient needs supplementary nutrition).
OMDQ MTS question 2 (Q2) score | Day 56 after completion or termination of radiotherapy
  Oral Mucositis Daily Questionnaire (OMDQ) mouth and throat soreness (MTS) question 2 (Q2) is a 5-point categorical scale in which patients grade MTS from 0 (no soreness) to 4 (extreme soreness)3 which is a component of the OMDQ in that it tracks very well with objective (WHO score and opioid use) and subjective measurement of OM severity.
OMAS | Day 56 after completion or termination of radiotherapy
  Oral Mucositis Assessment Scale (OMAS) provides an objective assessment of oral mucositis based on assessment of the appearance and extent of redness and ulceration in various areas of the mouth.